CLINICAL TRIAL: NCT02904330
Title: K1-70 - A Phase I, Single Ascending Intramuscular Dose or Single Ascending Intravenous Dose, Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study in Subjects With Graves' Disease
Brief Title: K1-70 - A Study in Subjects With Graves' Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AV7 Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K1im001
Record Dates: First submitted 2016-08-18; First posted 2016-09-16 (Estimated); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Graves' Disease
MeSH Terms: conditions — Graves Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single dose (Experimental): The intervention is K1-70 intramuscular or K1-70 intravenous. This is a single, ascending, intramuscular or intravenous dose, sequential group study.
  Interventions: Drug: K1-70 intramuscular or K1-70 intravenous

INTERVENTIONS:
Drug: K1-70 intramuscular or K1-70 intravenous — Each subject will receive one dose of K1-70 by IM injection or one dose of K1-70 by IV infusion on the morning of Day 1.

SUMMARY:
This study is the first time that K1-70 will be administered to humans. The principal aim of this study is to obtain safety and tolerability data when K1-70 is administered as an IM injection or as an IV infusion to subjects with Graves' disease.

Current therapy for Graves' disease includes treatment with anti-thyroid drugs, destruction of the thyroid using radioiodine, or total surgical thyroidectomy. Beta-blockers and calcium antagonists may be used to control some of the symptoms of hyperthyroidism.

K1-70 is a thyroid stimulating hormone receptor antagonist that may provide new in vivo diagnostic and therapeutic tools for the management of patients with Graves' disease, patients with thyroid cancer and patients who would benefit from controlling receptor activity.

DETAILED DESCRIPTION:
Graves' disease is one of the most common overt autoimmune disorders. Patients with Graves' disease have thyroid over activity and hyperthyroidism. Symptoms of hyperthyroidism include goitre, fatigue, heat intolerance, sweating, weight loss despite good appetite, shakiness, inappropriate anxiety, palpitations of the heart, shortness of breath, tetchiness and agitation, poor sleep, thirst, nausea and increased frequency of defaecation.

The rationale of this study is to obtain safety and tolerability data when K1-70 is administered as an intramuscular injection or as an IV infusion to subjects with Graves' disease.

This information, together with the pharmacokinetic data, will help establish the doses and dosage regimen suitable for repeat administration to patients.

This is an open-label study. The expected duration of each subject's participation in the study is approximately 18 weeks (including a screening period of up to 4 weeks).

ELIGIBILITY:
Main Inclusion Criteria:

* age 18-75 years
* have Graves' disease and are being treated with anti-thyroid medications OR not treated with anti-thyroid medications (due to side-effects) and who are clinically and biochemically euthyroid or hyperthyroid
* have a body mass index (weight [kg]/height [m]2) between 18.5 and 35.0 kg/m2

Main Exclusion Criteria:

* current or chronic history of liver disease
* history of cancer within the last 5 years except localised skin cancer
* Graves' orbitopathy with clinical activity score >3/7
* evidence of optic neuropathy and/or corneal breakdown
* significant systemic infection
* history of recurrent or current infection
* splenectomy
* recently had major surgery or plan major surgery
* had thromboembolic event due to a blood clot in the last 12 months
* have clinically significant laboratory tests
* a clinically significant allergic condition (excluding hay fever)
* currently receiving corticosteroids
* smoke more than 10 cigarettes (or its equivalent in nicotine (including use of e-cigarettes)) per day
* history of drug abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability will be measured using vital signs, ECG, blood samples for haematology, coagulation, clinical biochemistry and hormone panel, urinalysis, eye examinations, physical examinations and examination of injection or infusion site. | Over a period of 18 weeks
  Safety and tolerability testing consists of vital signs, ECG, blood samples for haematology, coagulation, clinical biochemistry and hormone panel, urine samples for urinalysis, eye examinations, physical examinations and examination of injection or infusion site. All clinically significant results and the number of treatment related adverse events will be reported.

SECONDARY OUTCOMES:
The concentration of K1-70 drug in the blood will be measured over time. | Over a period of 18 weeks
  The terminal elimination rate constant will be calculated and reported
The concentration of K1-70 drug in the blood will be measured over time. | Over a period of 18 weeks
  The terminal elimination half life will be calculated and reported
The concentration of K1-70 drug in the blood will be measured over time. | Over a period of 18 weeks
  Time of the maximum observed plasma concentration will be calculated and reported
The concentration of K1-70 drug in the blood will be measured over time. | Over a period of 18 weeks
  Maximum observed plasma concentration will be calculated and reported
The concentration of K1-70 drug in the blood will be measured over time. | Over a period of 18 weeks
  Area under the plasma concentration time curve to the last quantified concentration will be calculated and reported
The concentration of K1-70 drug in the blood will be measured over time. | Over a period of 18 weeks
  Area under the plasma concentration time curve from time zero to infinity will be calculated and reported
The concentration of K1-70 drug in the blood will be measured over time. | Over a period of 18 weeks
  Percentage of area under the plasma concentration time curve that is extrapolated will be calculated and reported
The antidrug antibodies will be measured to evaluate the immunogenic potential of K1-70 in Graves' disease patients | Over a period of 18 weeks
  The level of antidrug antibodies present in the patient serum will be measured over time and reported.
The effect of a single IM dose or single IV dose of K1-70 on thyroid activity in subjects with Graves' will be measured over time | Over a period of 18 weeks
  TSH levels will be measured and reported over time.
The effect of a single IM dose or single IV dose of K1-70 on thyroid activity in subjects with Graves' will be measured over time | Over a period of 18 weeks
  Free T3 levels will be measured and reported over time.
The effect of a single IM dose or single IV dose of K1-70 on thyroid activity in subjects with Graves' will be measured over time | Over a period of 18 weeks
  Free T4 levels will be measured and reported over time.

OTHER OUTCOMES:
Exploratory Objective: Thyroid hormones will be measured over time and their correlation to baseline TSH receptor autoantibody (TRAb) levels will be reported at different time points | Over a period of 18 weeks
  TSH levels will be reported against baseline TRAb over time.
Exploratory Objective: Thyroid hormones will be measured over time and their correlation to baseline TSH receptor autoantibody (TRAb) levels will be reported at different time points | Over a period of 18 weeks
  Free T3 levels will be reported against baseline TRAb over time.
Exploratory Objective: Thyroid hormones will be measured over time and their correlation to baseline TSH receptor autoantibody (TRAb) levels will be reported at different time points | Over a period of 18 weeks
  Free T4 levels will be reported against baseline TRAb over time.
Exploratory Objective: The potential effect of K1-70 on Graves' ophthalmopathy will be measured by eye examinations using the Clinical Activity Score (CAS) system. | Over a period of 18 weeks
  All clinically significant results and the number of treatment related adverse events will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, Professor, Principal Investigator — Medicines Evaluation Unit, Manchester, UK
Locations (2):
- United Kingdom (2):
  - Royal Liverpool University Hospital Clinical Research Unit, Liverpool
  - Medicines Evaluation Unit, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Evans M, Sanders J, Tagami T, Sanders P, Young S, Roberts E, Wilmot J, Hu X, Kabelis K, Clark J, Holl S, Richards T, Collyer A, Furmaniak J, Smith BR. Monoclonal autoantibodies to the TSH receptor, one with stimulating activity and one with blocking activity, obtained from the same blood sample. Clin Endocrinol (Oxf). 2010 Sep;73(3):404-12. doi: 10.1111/j.1365-2265.2010.03831.x. Epub 2010 Jun 9. PMID 20550534
- [Background] Sanders P, Young S, Sanders J, Kabelis K, Baker S, Sullivan A, Evans M, Clark J, Wilmot J, Hu X, Roberts E, Powell M, Nunez Miguel R, Furmaniak J, Rees Smith B. Crystal structure of the TSH receptor (TSHR) bound to a blocking-type TSHR autoantibody. J Mol Endocrinol. 2011 Feb 15;46(2):81-99. doi: 10.1530/JME-10-0127. Print 2011 Apr. PMID 21247981
- [Background] Furmaniak J, Sanders J, Young S, Kabelis K, Sanders P, Evans M, Clark J, Wilmot J, Rees Smith B. In vivo effects of a human thyroid-stimulating monoclonal autoantibody (M22) and a human thyroid-blocking autoantibody (K1-70). Auto Immun Highlights. 2011 Sep 14;3(1):19-25. doi: 10.1007/s13317-011-0025-9. eCollection 2012 Apr. PMID 26000124